CLINICAL TRIAL: NCT01578551
Title: A Randomized Phase II Study of Metformin Plus Paclitaxel/Carboplatin/Bevacizumab in Patients With Previously Untreated Advanced/Metastatic Pulmonary Adenocarcinoma
Brief Title: Study of Metformin Plus Paclitaxel/Carboplatin/Bevacizumab in Patients With Adenocarcinoma.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1188; NA_00052073 (Other: JHM IRB); 2P50CA058184-16 (NIH)
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Results first posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Adenocarcinoma
Keywords: Carcinoma, Non-Small-Cell Lung; Lung adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Paclitaxel; Carboplatin; Bevacizumab; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Paclitaxel, Carboplatin, Bevacizumab, and Metformin. Metformin starting at a dose of 500 mg twice a day, orally with meals. After one week, increase the dose of metformin to 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin treatment will be initiated one week before beginning chemotherapy, if possible, but chemotherapy will not be delayed for metformin loading.
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Bevacizumab; Drug: Metformin
- Arm B (Active Comparator): Paclitaxel, Carboplatin, and Bevacizumab
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel — 200 mg/m² IV over 3 hours, day 1 of each cycle. Paclitaxel + Carboplatin + Bevacizumab will be administered once every 21 days (Day 1) for up to 6 cycles. If subject has complete response, partial response, stable disease, or unacceptable toxicity. Bevacizumab with Metformin (Arm A) or Bevacizumab alone (Arm B) may continue as maintenance therapy.
  Other Names: Taxol; NSC 673089
Drug: Carboplatin — Carboplatin is administered at AUC= 6 mg/ml X min IV over 15-30 minutes, immediately following Paclitaxel infusion every 21 days
  Paclitaxel + Carboplatin + Bevacizumab will be administered once every 21 days (Day 1) for up to 6 cycles. If subject has complete response, partial response, stable disease, or unacceptable toxicity. Bevacizumab with Metformin (Arm A) or Bevacizumab alone (Arm B) may continue as maintenance therapy
  Other Names: platinum diamine; Paraplatin
Drug: Bevacizumab — All patients will receive the drug at 15 mg/kg every 21 days, given immediately after completion of chemotherapy, starting with Cycle 1. After induction chemotherapy is completed (4 cycles), bevacizumab will continue at 15 mg/kg every 21 days until PD (provided neither PD nor toxicity requiring discontinuation has occurred) measured from date of first dose of bevacizumab.
  Other Names: NSC 704865; RhuMAb VEGF; Recombinant Humanized Monoclonal Anti-VEGF Antibody
Drug: Metformin — 1000 mg twice daily with food.
  Other Names: N,N - dimethyl biguanide hydrochloride; glucophage
  Arms: Arm A

SUMMARY:
To determine the 1 year progression-free survival (PFS) of the combination of metformin and standard chemotherapy in patients with previously untreated advanced or metastatic pulmonary adenocarcinoma.

DETAILED DESCRIPTION:
Primary Objectives

To determine the 1 year progression-free survival (PFS) of the combination of metformin and standard chemotherapy in patients with previously untreated advanced or metastatic pulmonary adenocarcinoma.

Secondary Objectives

A. To evaluate the response to therapy and overall survival of the combination of metformin with standard chemotherapy in patients with previously untreated advanced or metastatic pulmonary adenocarcinoma.

B. To determine whether LKB1 gene status in tumors is a significant determinant of response when metformin is added to the therapy C. To acquire preliminary data regarding the effects of metformin on uptake of fluorodeoxyglucose in tumor and normal tissues.

Treatment will be administered on an outpatient basis.

Induction Therapy (Step 1, Cycles 1-4)

Metformin starting at a dose of 500 mg twice a day, orally with meals. After one week, increase the dose of metformin to 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin treatment will be initiated one week before beginning chemotherapy, if possible, but chemotherapy will not be delayed for metformin loading.

Paclitaxel 200 mg/m2 IV over 3 hours. For Paclitaxel pre-medication information

Carboplatin AUC = 6 mg/ml IV over 15 - 30 minutes, immediately following paclitaxel infusion

Bevacizumab 15 mg/kg IV infusion over 30 - 90 minutes

Metformin will be administered continuously, beginning one week before beginning chemotherapy, if possible, but chemotherapy will not be delayed for metformin loading. The other three drugs (paclitaxel, carboplatin, and bevacizumab) will be administered on day 1 of each 21 day cycle.

Maintenance Therapy

Patients responding to this therapy will be maintained with metformin (1000 mg twice daily) and bevacizumab (15 mg/kg IV over 30-90 minutes on day 1 of each 21-day cycle).

Duration of Therapy

In the absence of treatment delays due to adverse events, treatment may continue until one of the following criteria applies:

1. Disease progression,
2. Intercurrent illness that prevents further administration of treatment,
3. Unacceptable adverse events(s),
4. Patient decides to withdraw from the study, or
5. General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

ELIGIBILITY:
Inclusion Criteria:

Patients must have Histologically or cytologically confirmed non-squamous cell, non small cell carcinoma of the lung.

Patient must have measurable stage IV disease (includes M1a, M1b stages or recurrent disease) (according to the 7th edition of the TNM classification system). However, patients with T4NX disease (stage III B) with nodule(s) in ipsilateral lung lobe are not eligible, because such patients were not included in historical controls.

Patients be age >18 years.

Patients must have a Life Expectancy of greater than 12 weeks.

Patients must have an ECOG performance status 0 or 1 (Karnofsky > 70%; see Appendix A).

Patients must have normal organ and marrow function as defined below, within one week prior to randomization:

* absolute neutrophil count >1,500/mcL
* platelets > 100,000/mcL
* total bilirubin: within normal institutional limits
* AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
* creatinine ≤ 1.5 X institutional upper limit of normal
* urine dipstick for proteinuria of < less than 1+. If urine dipstick is > 1+ then a 24 hour urine for protein must demonstrate < 500 mg of protein in 24 hours to allow participation in the study.

Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Patients must have an INR < 1.5 and a PTT no greater than upper limits of normal within 1 week prior to randomization.

Patients with a history of hypertension must be well-controlled (<150sytolic/<100diastolic) on a stable regimen of anti-hypertensive therapy.

Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Patients with a history of gross hemoptysis (defined as bright red blood of ½ teaspoon or more) will be excluded from this trial.

Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.

Patients with a history of thrombotic or hemorrhagic disorders.

Patients receiving chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory agents known to inhibit platelet function. Treatment with dipyridamole (Persantine), ticlopidine (Ticlid), clopidogrel (Plavix) and/or cilostazol (Pletal)is also not allowed.

Patients receiving therapeutic anticoagulation. Prophylactic anticoagulation of venous access devices is allowed provided Section 3.10 is met. Caution should be taken on treating patients with low dose heparin or low molecular weight heparin for DVT prophylaxis during treatment with bevacizumab as there may be an increased risk of bleeding.

Prior use of chemotherapy.

Patients receiving immunotherapy, hormonal-therapy and or radiotherapy within 2 weeks prior to entering the study. Note: Those who have not recovered from adverse events due to these agents administered will be considered ineligible.

Patients receiving any other investigational agents.

Patients with a serious non-healing wound ulcer, or bone fracture, or major surgical procedure within 21 days prior to starting treatment.

Patients with uncontrolled brain metastasis. Note: Patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.

Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to metformin and paclitaxel or other agents used in the study are excluded.

Women that are pregnant or breastfeeding Note: Pregnant women are excluded from this study because the agents used in this study may be teratogenic to a fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with paclitaxel, breastfeeding women are also excluded from this study.

Patients that are HIV-positive on combination antiretroviral therapy due to the potential for lethal infections when treated with marrow-suppressive therapy.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ettinger, MD, Principal Investigator — Johns Hopkins SKCCC
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Johns Hopkins University SKCCC, Baltimore, Maryland

REFERENCES:
- [Result] Marrone KA, Zhou X, Forde PM, Purtell M, Brahmer JR, Hann CL, Kelly RJ, Coleman B, Gabrielson E, Rosner GL, Ettinger DS. A Randomized Phase II Study of Metformin plus Paclitaxel/Carboplatin/Bevacizumab in Patients with Chemotherapy-Naive Advanced or Metastatic Nonsquamous Non-Small Cell Lung Cancer. Oncologist. 2018 Jul;23(7):859-865. doi: 10.1634/theoncologist.2017-0465. Epub 2018 Feb 27. PMID 29487223

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Metformin dose of 500 mg twice a day After one week, increase dose of metformin to 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin tx initiated 1 week before beginning chemotherapy, chemotherapy not delayed for metformin loading.
  Paclitaxel: 200 mg/m² IV over 3 hours, day 1 of each cycle. Paclitaxel + Carboplatin + Bevacizumab will be administered once every 21 days (Day 1) for up to 6 cycles. If subject has complete response, partial response, stable disease, or unacceptable toxicity. Bevacizumab with Metformin (Arm A) or Bevacizumab alone (Arm B) may continue as maintenance therapy.
  Carboplatin: Carboplatin is administered at AUC= 6 mg/ml X min IV over 15-30 minutes, immediately following Paclitaxel infusion every 21 days
  Bevacizumab: 15 mg/kg every 21 days, every 21 days until PD
- Arm B: Paclitaxel: 200 mg/m² IV over 3 hours, day 1 of each cycle.
  Carboplatin: Carboplatin is administered at AUC= 6 mg/ml X min IV over 15-30 minutes, immediately following Paclitaxel infusion every 21 days
  Paclitaxel + Carboplatin + Bevacizumab will be administered once every 21 days (Day 1) for up to 6 cycles. If subject has complete response, partial response, stable disease, or unacceptable toxicity. Bevacizumab with Metformin (Arm A) or Bevacizumab alone (Arm B) may continue as maintenance therapy
  Bevacizumab: All patients will receive the drug at 15 mg/kg every 21 days, given immediately after completion of chemotherapy, starting with Cycle 1. After induction chemotherapy is completed (4 cycles), bevacizumab will continue at 15 mg/kg every 21 days until PD (provided neither PD nor toxicity requiring discontinuation has occurred) measured from date of first dose of bevacizumab.
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 19 | 6
Completed | 18 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Metformin starting at a dose of 500 mg twice a day, orally with meals. After one week, increase the dose of metformin to 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin treatment will be initiated one week before beginning chemotherapy, if possible, but chemotherapy will not be delayed for metformin loading.
  Paclitaxel: 200 mg/m² IV over 3 hours, day 1 of each cycle.
  .
  Carboplatin: Carboplatin is administered at AUC= 6 mg/ml X min IV over 15-30 minutes, immediately following Paclitaxel infusion every 21 days
  Paclitaxel + Carbop
- Arm B: Paclitaxel: 200 mg/m² IV over 3 hours, day 1 of each cycle. Paclitaxel + Carboplatin + Bevacizumab will be administered once every 21 days (Day 1) for up to 6 cycles. If subject has complete response, partial response, stable disease, or unacceptable toxicity. Bevacizumab with Metformin (Arm A) or Bevacizumab alone (Arm B) may continue as maintenance therapy.
  Carboplatin: Carboplatin is administered at AUC= 6 mg/ml X min IV over 15-30 minutes, immediately following Paclitaxel infusion every 21 days
  Paclitaxel + Carboplatin + Bevacizumab will be administered once every 21 days (Day 1) for up to 6 cycles. If subject has complete response, partial response, stable disease, or unacceptable toxicity. Bevacizumab with Metformin (Arm A) or Bevacizumab alone (Arm B) may continue as maintenance therapy
  Bevacizumab: All patients will receive the drug at 15 mg/kg every 21 days, given immediately after completion of chemotherapy, starting with
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 19 | 6 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 12 | 3 | 15
Age, Continuous [Median (Full Range); unit: years] | 58 [37 to 74] | 64 [55 to 70] | 61 [37 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 12 | 4 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 6 | 25

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Number of months without evidence of progression after 1 year of the combination of metformin and standard chemotherapy in patients with previously untreated advanced or metastatic pulmonary adenocarcinoma.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A: Metformin 500 mg twice a day, orally with meals. After one week, increase 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin treatment will be initiated one week before beginning chemotherapy, if possible, but chemotherapy will not be delayed for metformin loading.
  Paclitaxel: 200 mg/m² IV over 3 hours, day 1 of each cycle. Carboplatin: Carboplatin is administered at AUC= 6 mg/ml X min IV over 15-30 minutes, immediately following Paclitaxel infusion every 21 days
  Paclitaxel + Carboplatin + Bevacizumab will be administered once every 21 days (Day 1) for up to 6 cycles. If subject has complete response, partial response, stable disease, or unacceptable toxicity. Bevacizumab with Metformin (Arm A) or Bevacizumab alone (Arm B) may continue as maintenance therapy
  Bevacizumab: 15 mg/kg every 21 days, Metformin: 1000 mg twice daily with food.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 6
months | 9.6 [7.3 to NA] — The upper limits for the respective 95% confidence intervals could not be computed, given the small numbers of patients and censoring pattern. | 6.7 [4.4 to NA] — The upper limits for the respective 95% confidence intervals could not be computed, given the small numbers of patients and censoring pattern.

2. Secondary Outcome: Response to Therapy
Description: Percentage of participants with complete or partial response to combination of metformin with standard chemotherapy in patients with previously untreated advanced or metastatic pulmonary adenocarcinoma as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm A: Metformin starting at a dose of 500 mg twice a day, orally with meals. After one week, increase the dose of metformin to 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin treatment will be initiated one week before beginning chemotherapy, if possible, but chemotherapy will not be delayed for metformin loading.
  Paclitaxel: 200 mg/m² IV over 3 hours, day 1 of each cycle.
  Carboplatin: Carboplatin is administered at AUC= 6 mg/ml X min IV over 15-30 minutes, immediately following Paclitaxel infusion every 21 days
  Paclitaxel + Carboplatin + Bevacizumab will be administered once every 21 days (Day 1) for up to 6 cycles. If subject has complete response, partial response, stable disease, or unacceptable toxicity. Bevacizumab with Metformin (Arm A) or Bevacizumab alone (Arm B) may continue as maintenance therapy
  Bevacizumab: 15 mg/kg every 21 days,
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 6
percentage of participants | 56 [31 to 78] | 33 [6 to 76]

3. Secondary Outcome: Overall Survial
Description: Number of months alive after 1 year of the combination of metformin with standard chemotherapy in patients with previously untreated advanced or metastatic pulmonary adenocarcinoma.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 18 | 6
months | 15.9 [8.4 to NA] — The upper limits for the respective 95% confidence intervals could not be computed, given the small numbers of patients and censoring pattern. | 13.9 [12.7 to NA] — The upper limits for the respective 95% confidence intervals could not be computed, given the small numbers of patients and censoring pattern.

ADVERSE EVENTS:
Time Frame: up to 1 year
Groups:
- Arm A: Metformin starting at a dose of 500 mg twice a day, orally with meals. After one week, increase the dose of metformin to 1000 mg as the first dose of the day and 500 mg as the second dose. After another week, increase to 1000 mg of metformin two times a day. Metformin treatment will be initiated one week before beginning chemotherapy, if possible, but chemotherapy will not be delayed for metformin loading.
  Paclitaxel: 200 mg/m² IV over 3 hours, day 1 of each cycle.
  Carboplatin: Carboplatin is administered at AUC= 6 mg/ml X min IV over 15-30 minutes, immediately following Paclitaxel infusion every 21 days
  Bevacizumab: 15 mg/kg every 21 days, Metformin: 1000 mg twice daily with food.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/6
Other Adverse Events (participants affected / at risk) | 19/19 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=19) | Arm B (N=6)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=19) | Arm B (N=6)
White blood cell count decreased (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 10 (10) | 2 (2)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4 (4) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Catheter-related infection (Infections and infestations) | 1 (1) | 0 (0)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hypophosphatemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dehydration (Gastrointestinal disorders) | 2 (2) | 1 (1)
Infusion related reaction (Investigations) | 1 (1) | 2 (2)
Headache (Investigations) | 1 (1) | 0 (0)
Neuropathy (Investigations) | 0 (0) | 1 (1)
Arthralgia (General disorders) | 1 (1) | 0 (0)
Pain in extremity (General disorders) | 0 (0) | 1 (1)
Bone pain (General disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 3 (3) | 0 (0)
Thomboembolic event (Cardiac disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes